CLINICAL TRIAL: NCT03352193
Title: Specific Oral Tolerance Induction (SOTI) to Children With IgE-mediated Wheat Allergy
Status: Recruiting | Type: Observational
Sponsor: Athens General Children's Hospital "Pan. & Aglaia Kyriakou" (Other)
Responsible Party: Principal Investigator, Nikolaos Kitsioulis, MD, Athens General Children's Hospital "Pan. & Aglaia Kyriakou"
Other Study IDs: Wheat SOTI
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Wheat Allergy
MeSH Terms: conditions — Wheat Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum

GROUPS / COHORTS (2):
- SOTI group: Wheat spaghetti
  Interventions: Dietary Supplement: Wheat spaghetti
- Historical control group: No intervention

INTERVENTIONS:
Dietary Supplement: Wheat spaghetti — Wheat oral immunotherapy
  Groups: SOTI group

SUMMARY:
This is an observational pilot study investigating the effectiveness, safety and specific immunological mechanisms of Specific Oral Tolerance Induction (SOTI) in children with IgE-mediated wheat allergy.

The study will include 10 patients with persistent IgE-mediated allergy to wheat, who will undergo 1-year home SOTI. Moreover, 5 patients with IgE-mediated allergy to wheat will be followed for 1-year period after their diagnosis, without any intervention.

Well-cooked wheat spaghetti will be given daily to patients with a programmed weekly dose increment for 27 weeks (up-dosing phase).

Subsequently, wheat protein maintenance dose will be received daily for additional 6 months (maintenance phase), while afterwards patients will be clinically assessed and a 2nd OFC at a higher cumulative dose of wheat protein will be performed, in order to assess patients' desensitization to wheat.

Skin Prick Tests (SPTs) to wheat, blood sampling for the determination of total IgE, wheat specific IgEs and wheat Basophil Activation Test (BAT) will be performed at baseline, when patients reach the maintenance dose and before the 2nd OFC.

Regarding historical control group the same testing will be performed at baseline and at re-evaluation (post 12 months).

DETAILED DESCRIPTION:
This is an observational pilot study investigating the effectiveness, safety and specific immunological mechanisms of Specific Oral Tolerance Induction (SOTI) in children aged 2-16 years with IgE-mediated wheat allergy. The study will be conducted in the Department of Allergy and Clinical Immunology, 2nd University Pediatric Clinic of "Panagiotis & Aglaia Kyriakou" Children's Hospital, Athens, Greece.

The study will include 10 patients with persistent IgE-mediated allergy to wheat, who will undergo 1-year home SOTI, defined as SOTI group. Moreover, 5 patients with IgE-mediated allergy to wheat will be followed for 1-year period after their diagnosis, without any intervention, either because of denial or due to positive history of severe anaphylaxis to very low doses of wheat during baseline Oral Food Challenge / OFC or home ingestion in the preceding 3 months. These will be defined as historical control group.

Well-cooked wheat spaghetti will be given daily to patients with a programmed weekly dose increment for 27 weeks (up-dosing phase). Three different home starting doses will be pre-determined in accordance to each individual's reactivity threshold during baseline OFC to wheat. Each proposed starting dose will be associated with a different weekly stable increase ratio of wheat intake, so that all patients reach an equal predefined maintenance dose at week 27 of up-dosing phase.

Subsequently, wheat protein maintenance dose (spaghetti or equivalent quantity of wheat protein of other wheat product) will be received daily for additional 6 months (maintenance phase), while afterwards patients will be clinically assessed and a 2nd OFC at a higher cumulative dose of wheat protein will be performed, in order to assess patients' desensitization to wheat.

Skin Prick Tests (SPTs) to wheat, blood sampling for the determination of total IgE, wheat specific IgEs (f4, f79, f98, f416, f433) and wheat Basophil Activation Test (BAT) will be performed at baseline, when patients reach the maintenance dose and before the 2nd OFC. Additionally, blood sampling for determination of the levels of anti-tissue transglutaminase (tTG)-IgA/IgG and anti-endomysial (EMA)-IgA antibodies at baseline and post study completion will be performed.

Regarding historical control group the same testing (except anti-tTG and anti-EMA) will be performed at baseline visit and at re-evaluation (post 12 months). All children and / or their parents / legal guardians will be trained in the use of self-injectable epinephrine in case of severe allergic reactions and a detailed treatment plan will be given by the study doctors. Written information sheet will be provided and written consent will be obtained from all parents/legal guardians.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-16 years
2. Personal history of IgE-mediated allergy to wheat with unequivocal allergic reaction one year before study entry, and

   1. Positive SPT in wheat (> 3 mm), and/or
   2. Wheat specific IgE f4 > 0.35 kUa/L, and
   3. A positive Oral Food Challenge (OFC) to wheat, with the exception of patients who report a recent reaction (< 3 months before study entry) after the consumption of wheat products
3. Signed written consent form of the parents.

Exclusion Criteria:

1. Severe persistent or uncontrolled bronchial asthma or other lung disease (other than asthma), and/or
2. Recent personal history (over the past 12 months) of severe anaphylactic reaction following wheat consumption, for which Intensive Care Unit (ICU) hospitalization was required, and/or
3. Patients on specific immunotherapy, subcutaneous (SCIT) or sublingual (SLIT) or any other form of current immunotherapy or treatment with other biological agents, and/or
4. Personal history of anaphylaxis due to wheat-dependent exercise induced anaphylaxis, and/or
5. Patients with celiac disease or diagnosis other than IgE-mediated wheat allergy (eg eosinophilic gastrointestinal diseases), and/or
6. Patients with cardiovascular disease or other significant systemic disease, and/or
7. Patients presenting severe anaphylactic reaction to very low doses of wheat (eg. after administration of the 1st or 2nd dose during the baseline OFC).

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Wheat allergic patients visiting the Allergy Department of a tertiary University Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Wheat allergic children achieving desensitization after 1 year of wheat home SOTI. | 1 year
  The rate of wheat allergic children achieving desensitization after 1 year of wheat home SOTI.

SECONDARY OUTCOMES:
Variability of Skin Prick Tests (SPTs) pre and post 1-year SOTI intervention | 1 year
  Determination of Skin Prick Tests (SPTs) of wheat allergic children pre and post 1-year SOTI intervention
Total IgE, wheat specific IgE levels (f4, f79, f98, f416, f433) pre and post 1-year SOTI intervention | 1 year
  Determination of wheat allergic patients' total IgE, wheat specific IgE levels (f4, f79, f98, f416, f433) pre and post 1-year SOTI intervention
Wheat basophil activation test (BAT) pre and post 1-year SOTI intervention | 1 year
  Determination of wheat allergic patients' basophils activation pre and post 1-year SOTI intervention via Basophil Activation Test (BAT)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Kitsioulis, MD, Principal Investigator — National and Kapodistrian University of Athens; Nikolaos Papadopoulos, MD, PhD, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- Department of Allergy and Clinical Immunology, 2nd Pediatric Clinic, General Children's Hospital P-A Kyriakou, Athens, Greece